CLINICAL TRIAL: NCT00174174
Title: A Placebo Control, Double Blind, Cross Over Study of Modafinil in Patients With Narcolepsy
Brief Title: Provigil (Modafinil) Study by Taiwan Biotech Co.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 920203l
Record Dates: First submitted 2005-09-14; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-10

CONDITIONS: Narcolepsy; Cataplexy; Sleep Disorders; Hypersomnolence; Excessive Sleepiness
MeSH Terms: conditions — Narcolepsy; Cataplexy; Sleep Wake Disorders; Disorders of Excessive Somnolence | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The primary objective is to evaluate the therapeutic effect of excessive daytime sleepiness associated with narcolepsy. Both of the subjective and objective sleepiness of the patients were assessed in the experiment by repeat measures.

ELIGIBILITY:
Inclusion Criteria:

* Polysomnographic findings of shortened sleep latency less than 5 minutes average of Multiple Sleep Latency Test, and two or more SOREM should be fulfilled.
* Age of 12 y/o to 55 y/o.
* The liver and kidney functions are within normal limits.
* Meeting the strict criteria of narcolepsy described above.
* Wash out any medications which might enhance wakefulness or affect nocturnal sleep two weeks prior to the experiments.
* Willingness to comply with the protocol and signed the written Informed Consent.

Exclusion Criteria:

* Patients whose hypersomnia was caused by severely sleep deprived, phase delayed, or suspected long sleeper.
* Patients with concomitant neurological disorder and psychiatric disorders.
* Patients with sleep-related breathing disorders whose apnea/hypopnea index (AHI) was 5 pauses per hour above.
* Patients with Restless Leg Syndrome & Periodic Limbs Movements whose index was more than 5 per hour.
* Patients who are pregnant or breast-feeding.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-09

PRIMARY OUTCOMES:
The change from baseline in the sleep latency.

SECONDARY OUTCOMES:
Patient's assessment of general level of daytime sleepiness on ESS.
Patient's cognitive function assessed by psychomotor function test (Trail making test, and Digit Symbol Substitution Test).
Patient's sleep quality evaluated by PSQI.
Safety would be evaluated by tabulating and summarizing all adverse events reported.

CONTACTS AND LOCATIONS:
Overall Officials: Yue-Joe Lee, M.D., Principal Investigator — Department of Psychiatry, National Taiwan University